CLINICAL TRIAL: NCT05957237
Title: Evaluation of Characteristics of Patients With Nonsurgical Complications After Bariatric Surgery and Quality of Life in Patients Hospitalised in UZ Leuven
Brief Title: Evaluation of Characteristics of Patients With Nonsurgical Complications After Bariatric Surgery and Quality of Life
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s59712
Record Dates: First submitted 2022-06-10; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subjects hospitalised with non-surgical complications after bariatric surgery (case)
- Subjects with bariatric surgery without nonsurgical complications (control)
- Subjects with obesity (control)

SUMMARY:
Retrospective study: Analysis of characteristics of patients that were hospitalised with nonsurgical complications after bariatric surgery.

Cross-sectional study: To present and evaluate (clinical) parameters and quality of life measures of patients with nonsurgical complications after bariatric surgery compared to bariatric patients without hospitalisation for complications and obese patients.

DETAILED DESCRIPTION:
Retrospective study: The general objective is to describe and evaluate the characteristics of patients with nonsurgical complications after bariatric surgery based on parameters registered in the medical record.

Cross-sectional study:

1. Primary objective: To evaluate how quality of life is perceived in patients hospitalised for nonsurgical complications after bariatric surgery compared to control groups through Health-related Quality of Life (HRQoL) questionnaires.
2. Secondary objectives: To evaluate and compare (clinical) parameters and scoring on questionnaires about impact of weight, physical activity, anxiety and depression, impulsivity, alcohol use and eating behaviour for different bariatric and obese populations.

ELIGIBILITY:
CROSS-SECTIONAL STUDY

Patients hospitalised with non-surgical complications of bariatric surgery

* Inclusion Criteria:

  * Signed informed consent
  * Patients underwent bariatric surgery
  * Patients are hospitalised for nonsurgical complications of bariatric surgery at the Endocrinology unit of UZ Leuven
* Exclusion Criteria:

  * Patients are not able to complete the questionnaires themselves
  * Patients who do not understand Dutch

Patients with bariatric surgery who were never hospitalised with non-surgical complications

* Inclusion Criteria:

  * Signed informed consent
  * Patients underwent bariatric surgery
  * Patients without history of hospitalisation for nonsurgical complications of bariatric surgery
* Exclusion Criteria:

  * Patients are not able to complete the questionnaires themselves
  * Patients who do not understand Dutch

Patients with obesity

* Inclusion Criteria:

  * Signed informed consent
  * Patients visit the Obesity Clinic of UZ Leuven
* Exclusion Criteria:

  * Patients are not able to complete the questionnaires themselves
  * Patients who do not understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised with non-surgical complications of bariatric surgery Patients with bariatric surgery who were never hospitalised with non-surgical complications Patients with obesity
Sampling Method: Probability Sample
Enrollment: 796 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
RETROSPECTIVE STUDY: Type of non-surgical complication | 01/01/2014 to 31/12/2018
  Collect the type of non-surgical complication following bariatric surgery for which the patient is hospitalised
CROSS-SECTIONAL STUDY: Quality of life | Moment of inclusion
  Using the WHODAS 2.0 questionnaire, health-related quality of life will be assessed.

SECONDARY OUTCOMES:
CROSS-SECTIONAL STUDY: Scores on questionnaire concerning impact of weight | Questionnaires are to be completed at the moment of inclusion
  IWQOL-Lite
CROSS-SECTIONAL STUDY: Scores on questionnaires concerning physical activity | Questionnaires are to be completed at the moment of inclusion
  IPAQ
CROSS-SECTIONAL STUDY: Scores on questionnaires concerning anxiety, depression and personality disorders | Questionnaires are to be completed at the moment of inclusion
  CIDI
CROSS-SECTIONAL STUDY: Scores on questionnaires concerning impulsivity | Questionnaires are to be completed at the moment of inclusion
  BIS-11
CROSS-SECTIONAL STUDY: Scores on questionnaires concerning alcohol use | Questionnaires are to be completed at the moment of inclusion
  AUDIT
CROSS-SECTIONAL STUDY: Scores on questionnaires concerning eating behaviour | Questionnaires are to be completed at the moment of inclusion
  EDE-Q
CROSS-SECTIONAL STUDY: Scores on questionnaires concerning eating behaviour | Questionnaires are to be completed at the moment of inclusion
  eating behaviour after bariatric surgery (questionnaire developed at UZ Leuven)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mertens, MD PhD, Principal Investigator — UZ Leuven

IPD SHARING:
Plan to Share IPD: Undecided